CLINICAL TRIAL: NCT01216072
Title: A 6-month, Randomized, Active Comparator, Open-label, Multi-Center Study to Evaluate Patient OutComes, Safety and Tolerability of Fingolimod (FTY720) 0.5 mg/Day in Patients With Relapsing Forms of Multiple Sclerosis Who Are Candidates for MS Therapy Change From Previous Disease Modifying Therapy (EPOC)
Brief Title: A 6-month, Randomized, Open-label, Patient OutComes, Safety and Tolerability Study of Fingolimod (FTY720) 0.5 mg/Day vs. Comparator in Patients With Relapsing Forms of Multiple Sclerosis
Acronym: EPOC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720DUS01
Record Dates: First submitted 2010-09-07; First posted 2010-10-07 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Relapsing Forms of Multiple Sclerosis
Keywords: Relapsing Forms of Multiple Sclerosis; Disease Modifying Therapy; fingolimod; Patient Reported Outcomes
MeSH Terms: interventions — Fingolimod Hydrochloride; Interferon beta-1a; Glatiramer Acetate; Interferon beta-1b

ARMS (2):
- Fingolimod (Experimental): Patients randomized in this arm received Fingolimod 0.5 mg/day oral capsule for 6 months core period .
  Interventions: Drug: Fingolimod
- Multiple Sclerosis Disease Modifying Treatments (MS DMTs) (Active Comparator): Patients randomized in this arm received selected Standard MS DMT such as Interferon beta-1b or Interferon beta-1a or Glatiramer acetate for 6 months. An open-label extension of up to 3 months of treatment with fingolimod was to be available for patients in the DMT arm who successfully completed all study visits.
  Interventions: Drug: Standard MS DMTs

INTERVENTIONS:
Drug: Fingolimod — 0.5 mg/day oral capsule
  Other Names: GILENYA™
  Arms: Fingolimod
Drug: Standard MS DMTs
  Other Names: Avonex®,; Copaxone®,; Rebif®,; Betaseron®,; Extavia®
  Arms: Multiple Sclerosis Disease Modifying Treatments (MS DMTs)

SUMMARY:
The purpose of this study is to evaluate the change in patient-reported outcomes, physician assessment of a change as well as safety and tolerability in patients with Relapsing Forms of Multiple Sclerosis on previous Disease Modifying Therapy (DMT) who are randomized to one of two treatment arms: fingolimod vs. standard of care DMT.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing forms of MS
* Expanded Disability Status Scale (EDSS) 0-5.5
* Continuous treatment with MS DMT for a minimum of 6 months
* Fingolimod naive

Exclusion Criteria:

* Immune system diseases other than MS
* Active macular edema
* History of selected prior infections and criteria for immunizations
* History of selected immune system treatments and/or medications
* Selected cardiovascular, pulmonary, or hepatic conditions
* Selected abnormal laboratory values
* Pregnant or nursing women

Other protocol-defined inclusion/exclusion criteria applied

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (134):
- United States (128):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Cullman, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Berkeley, California
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, La Habra, California
  - Novartis Investigative Site, Loma Linda, California
  - Novartis Investigative Site, Newport Beach, California
  - Novartis Investigative Site, Oceanside, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Boulder, Colorado
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Fort Collins, Colorado
  - Novartis Investigative Site, Fairfield, Connecticut
  - Novartis Investigative Site, New London, Connecticut
  - Novartis Investigative Site, Stratford, Connecticut
  - Novartis Investigative Site, Dover, Delaware
  - Novartis Investigative Site, Newark, Delaware
  - Novartis Investigative Site, Atlantis, Florida
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Doral, Florida
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Lighthouse PT, Florida
  - Novartis Investigative Site, Maitland, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Pompano Beach, Florida
  - Novartis Investigative Site, Ponte Vedra Beach, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Sunrise, Florida
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Vero Beach, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Columbus, Georgia
  - Novartis Investigative Site, Decatur, Georgia
  - Novartis Investigative Site, Idaho Falls, Idaho
  - Novartis Investigative Site, Elk Grove Village, Illinois
  - Novartis Investigative Site, Evanston, Illinois
  - Novartis Investigative Site, Flossmoor, Illinois
  - Novartis Investigative Site, Northbrook, Illinois
  - Novartis Investigative Site, Anderson, Indiana
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Merrillville, Indiana
  - Novartis Investigative Site, Valparaiso, Indiana
  - Novartis Investigative Site, Des Moines, Iowa
  - Novartis Investigative Site, Lenexa, Kansas
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Destrehan, Louisiana
  - Novartis Investigative Site, Hammond, Louisiana
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, Shreveport, Louisiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Bethesda, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Springfield, Massachusetts
  - Novartis Investigative Site, Worcester, Massachusetts
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Grand Rapids, Michigan
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Novartis Investigative Site, Southfield, Michigan
  - Novartis Investigative Site, Bolivar, Missouri
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Nixa, Missouri
  - Novartis Investigative Site, North Kansas City, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Billings, Montana
  - Novartis Investigative Site, Freehold, New Jersey
  - Novartis Investigative Site, Somerset, New Jersey
  - Novartis Investigative Site, Teaneck, New Jersey
  - Novartis Investigative Site, Toms River, New Jersey
  - Novartis Investigative Site, Amherst, New York
  - Novartis Investigative Site, Latham, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Patchogue, New York
  - Novartis Investigative Site, Plainview, New York
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Burlington, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Greenville, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Salisbury, North Carolina
  - Novartis Investigative Site, Wilmington, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Akron, Ohio
  - Novartis Investigative Site, Bellevue, Ohio
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Uniontown, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Corvallis, Oregon
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Monroeville, Pennsylvania
  - Novartis Investigative Site, Rumford, Rhode Island
  - Novartis Investigative Site, Beufort, South Carolina
  - Novartis Investigative Site, Columbia, Tennessee
  - Novartis Investigative Site, Cordova, Tennessee
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Colleyville, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Lubbock, Texas
  - Novartis Investigative Site, Plano, Texas
  - Novartis Investigative Site, Round Rock, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Sherman, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Newport News, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Roanoke, Virginia
  - Novartis Investigative Site, Vienna, Virginia
  - Novartis Investigative Site, Kirkland, Washington
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Morgantown, West Virginia
- Canada (5):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Nepean, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Guaynabo, Puerto Rico

REFERENCES:
- [Derived] Hughes B, Cascione M, Freedman MS, Agius M, Kantor D, Gudesblatt M, Goldstick LP, Agashivala N, Schofield L, McCague K, Hashmonay R, Barbato L; EPOC study investigators. First-dose effects of fingolimod after switching from injectable therapies in the randomized, open-label, multicenter, Evaluate Patient OutComes (EPOC) study in relapsing multiple sclerosis. Mult Scler Relat Disord. 2014 Sep;3(5):620-8. doi: 10.1016/j.msard.2014.06.006. Epub 2014 Jul 3. PMID 26265274
- [Derived] Fox E, Edwards K, Burch G, Wynn DR, LaGanke C, Crayton H, Hunter SF, Huffman C, Kim E, Pestreich L, McCague K, Barbato L; EPOC study investigators. Outcomes of switching directly to oral fingolimod from injectable therapies: Results of the randomized, open-label, multicenter, Evaluate Patient OutComes (EPOC) study in relapsing multiple sclerosis. Mult Scler Relat Disord. 2014 Sep;3(5):607-19. doi: 10.1016/j.msard.2014.06.005. Epub 2014 Jul 4. PMID 26265273
- [Derived] Calkwood J, Cree B, Crayton H, Kantor D, Steingo B, Barbato L, Hashmonay R, Agashivala N, McCague K, Tenenbaum N, Edwards K. Impact of a switch to fingolimod versus staying on glatiramer acetate or beta interferons on patient- and physician-reported outcomes in relapsing multiple sclerosis: post hoc analyses of the EPOC trial. BMC Neurol. 2014 Nov 26;14:220. doi: 10.1186/s12883-014-0220-1. PMID 25424122
- [Derived] Cascione M, Wynn D, Barbato LM, Pestreich L, Schofield L, McCague K. Randomized, open-label study to evaluate patient-reported outcomes with fingolimod after changing from prior disease-modifying therapy for relapsing multiple sclerosis: EPOC study rationale and design. J Med Econ. 2013 Jul;16(7):859-65. doi: 10.3111/13696998.2013.802239. Epub 2013 May 20. PMID 23647445
- See also: Click here for more information about this study: — http://www.NovartisClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients randomized in a 3:1 ratio to either fingolimod (0.5 mg/day) or MS DMT.
Groups:
- Fingolimod: Patients randomized in this arm received Fingolimod 0.5 mg/day oral capsule for 6 months core period.
Period: Open-Label Core Period ( 6 Months)
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatments (MS DMTs)
Started | 790 | 263
Full Analysis Set | 789 (One patient was randomized in error and was not included in FAS.) | 263
Safety Set | 783 | 245
Completed | 714 | 229
Not Completed | 76 | 34
Not completed — Adverse Event | 40 | 4
Not completed — Abnormal laboratory value(s) | 2 | 0
Not completed — Abnormal test procedure result(s) | 3 | 0
Not completed — Lack of Efficacy | 3 | 4
Not completed — Withdrawal by Subject | 12 | 22
Not completed — Lost to Follow-up | 5 | 0
Not completed — Protocol Deviation | 11 | 4
Period: Open-Label Extension Period (3 Months)
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatments (MS DMTs)
Started | 0 | 195 (Only DMT patients, who completed the core study, were eligible for fingolimod.)
Safety Set | 0 | 193
Completed | 0 | 181
Not Completed | 0 | 14
Not completed — Adverse Event | 0 | 10
Not completed — Abnormal test procedure results | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatments (MS DMTs) | Total
Number analyzed (Participants) | 790 | 263 | 1053
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (9.82) | 45.1 (9.82) | 45.8 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 601 | 208 | 809
  Male | 189 | 55 | 244

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Global Satisfaction Subscale of the Treatment Satisfaction Questionnaire for Medication (TSQM) at Month 6
Description: The TSQM was developed and validated as a general measure for treatment satisfaction. It contains 14 items assessing the following 4 domains: effectiveness (sum of scores for questions 1 - 3), side effects (sum of scores for questions 4 - 8), convenience (sum of scores for questions 9 - 11) and Global Satisfaction (sum of scores for questions 12 - 14). The primary analysis was on Global Satisfaction. Question 12 scored as 1(not at all confident) to 5 (extremely confident); question 13 scored as 1(not at all certain) to 5(extremely certain); and question 14 scored as 1(extremely dissatisfied) to 7(extremely satisfied). The scores of the domain were added together and an algorithm was used to create a score of 0 to 100. Higher scores indicated greater satisfaction. A positive change from baseline indicates improvement.
Time Frame: Baseline, Month 6
Population: This analysis was conducted using the Full Analysis Set. The Full Analysis Set comprised all randomized patients to whom study medication was assigned. Patients with both baseline and 6 month assessments were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatments (MS DMTs)
Number analyzed (Participants) | 714 | 221
units on a scale | 22.5 (27.1) | 3.5 (20.57)

2. Secondary Outcome: Number of Patients Who Experienced Adverse Events, Serious Adverse Events and Death
Description: In this analysis, patients with all (serious and non-serious) adverse events, serious adverse events and death were reported.
Time Frame: 9 months (6 month core + 3 month Extension)
Population: Safety Set included all patients who received at least one dose of study drug.
Measure: Number; unit: Participants
Groups:
- Multiple Sclerosis Disease Modifying Treatments (MS DMTs): Patients randomized in this arm received selected Standard MS DMT such as Interferon beta-1b or Interferon beta-1a or Glatiramer acetate for 6 months.
- Extension Fingolimod Period: An open-label extension of up to 3 months of treatment with fingolimod was to be available for patients in the DMT arm who successfully completed all study visits.
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatments (MS DMTs) | Extension Fingolimod Period
Number analyzed (Participants) | 783 | 245 | 193
Participants
  Adverse Events (serious and non-serious) | 617 | 152 | 123
  Serious Adverse Events | 31 | 5 | 7
  Death | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Patient-reported Activities of Daily Living (ADL) Using the Multiple Sclerosis Activities Scale (PRIMUS-Activities) at Month 6
Description: The PRIMUS activity measure is a 15-item assessment of patient-reported ADL. The PRIMUS-Activities total score was calculated by summing the 15 item scores after recoding the responses from 1 - 3 to 0 - 2. Totals scores range from 0 to 30 with higher scores indicating greater activity limitation. If no more than 20% of the items were missing, the total score was the product of the mean response of the non-missing items and the total number of items. If more than 20% of all items were missing, the total score was set to missing. A negative change from baseline indicates improvement.
Time Frame: Baseline, Month 6
Population: This analysis was conducted using the Full Analysis Set. The Full Analysis Set comprised all randomized patients to whom study medication was assigned. Patients with both baseline and 6 month assessments were included in this analysis. Missing values were imputed using the Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatments (MS DMTs)
Number analyzed (Participants) | 734 | 234
units on a scale | -0.6 (4.51) | -0.2 (4.97)

4. Secondary Outcome: Change From Baseline in Patient-reported Fatigue Using the Fatigue Severity Scale (FSS)
Description: The Fatigue Severity Scale (FSS) is a 9-item assessment scale measuring fatigue and its effects, using a scale from 1 to 7, with higher scores indicating greater fatigue, or greater negative effects of fatigue on daily living. The FSS 9 item total score was calculated by summing the first 9 item scores and dividing by the number of non-missing items. If no more than 20% of the items were missing, the total score was the product of the mean response of the non missing items and the total number of items. If more than 20% of all items were missing, the total score was set to missing. A negative change from baseline indicates improvement.
Time Frame: Baseline, Month 3, Month 6
Population: This analysis was conducted using the Full Analysis Set. The Full Analysis Set comprised all randomized patients to whom study medication was assigned. Patients with baseline to 3 month assessments and/or baseline to 6 month assessments were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatments (MS DMTs)
Number analyzed (Participants) | 789 | 263
units on a scale
  Change from Baseline to Month 3 (n=710,232) | -0.3 (1.24) | 0.0 (1.14)
  Change from Baseline to Month 6 (n=687,218) | -0.4 (1.24) | 0.0 (1.13)

5. Secondary Outcome: Change From Baseline in the Patient-reported Effectiveness Subscale Using the TSQM v1.4
Description: The effectiveness scale was scored as follows: 1(extremely dissatisfied) to 7(extremely satisfied). The scores of the domain were added together and an algorithm was used to create a score of 0 to 100. Higher scores indicated greater satisfaction. A positive change from baseline indicates improvement.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatments (MS DMTs)
Number analyzed (Participants) | 723 | 225
units on a scale | 15.5 (27.53) | 2.8 (19.05)

6. Secondary Outcome: Change From Baseline in the Patient-reported Side Effects Subscale Using the TSQM v1.4
Description: The Side Effects subscale was scored as follows: question 4 scored as 0(no) or 1(yes); question 5 scored as 1(extremely bothersome) to 5(not at all bothersome); and questions 6 - 8 scored as 1(a great deal) to 5(not at all). The scores of the domain were added together and an algorithm was used to create a score of 0 to 100. Higher scores indicated greater satisfaction. A positive change from baseline indicates improvement.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatments (MS DMTs)
Number analyzed (Participants) | 708 | 219
units on a scale | 22.9 (29.89) | 3.5 (23.18)

7. Secondary Outcome: Change From Baseline in the Patient-reported Convenience Subscale Using the TSQM v1.4
Description: The convenience subscale was scored as follows: questions 9 and 10 scored as 1(extremely difficult) to 7 (extremely easy), and question 11 scored as 1(extremely inconvenient) to 7 (extremely convenient). The scores of the domain were added together and an algorithm was used to create a score of 0 to 100. Higher scores indicated greater satisfaction. A positive change from baseline indicates improvement.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatments (MS DMTs)
Number analyzed (Participants) | 718 | 222
units on a scale | 41.8 (22.85) | 1.5 (18.33)

8. Secondary Outcome: Change From Baseline in Patient-reported Health-related Quality-of-life Using the Short Form Health Survey v2 Standard (SF-36 v2)
Description: The SF-36v2 is a validated health-related quality of life instrument used in numerous disease states, including MS. It is a self-administered survey that measures 8 domains of health including: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems and general mental health. Additionally, two summary scale scores can be calculated: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). If half or more questions within a domain were answered, then a score was calculated for that domain. Otherwise, the patient score for that domain was set to missing. If the patient was missing any 1 of the 8 scale scores, then the physical and mental component scores were set to missing. An algorithm was used to create a score from 0 to 100 for each domain score and component score. A positive change from baseline indicates improvement.
Time Frame: Baseline, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatments (MS DMTs)
Number analyzed (Participants) | 789 | 263
units on a scale
  Physical Function (n=745,226) | 1.5 (7.96) | 0.4 (7.03)
  Role Limitations d/t Physical Health (n=742,226) | 2.8 (9.65) | 1.2 (8.51)
  Bodily Pain (n=742,226) | 2.0 (9.7) | -0.3 (8.38)
  General Health Perceptions (n=737,224) | 0.8 (8.29) | -0.3 (7.24)
  Vitality (n=745,227) | 2.8 (8.88) | 0.6 (7.73)
  Social Functioning (n=747,227) | 2.6 (10.31) | 0.8 (10.61)
  Role Limitation d/t Emotional Problems (n=745,226) | 1.6 (12.48) | -0.6 (11.51)
  General Mental Health (n=745,227) | 2.2 (9.62) | 0.3 (9.37)
  Physical Component Summary Scale (n=724,222) | 1.7 (7.41) | 0.3 (6.48)
  Mental Component Summary Scale (n=724,222) | 2.3 (10.03) | 0.2 (9.62)

9. Secondary Outcome: Change From Baseline in Patient-reported Depression Using the Beck Depression Inventory (BDI-II)
Description: The Beck Depression Inventory (BDI-II) is a 21-question multiple-choice self-report inventory. Each item is scored from 0 to 3. The questions in the BDI-II refer to how the patient has been feeling over the past two weeks specifically. The BDI-II total score was calculated by summing the 21 item scores. Final scores ranged from 0 to 63 where higher scores indicated more severe depression. If no more than 20% of the items were missing, the total score was the product of the mean response of the non-missing items and the total number of items. If more than 20% of all items were missing, the total score was set to missing. A negative change indicates improvement.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatments (MS DMTs)
Number analyzed (Participants) | 789 | 263
units on a scale
  Change from Baseline to Month 3 (n=748,236) | -3.2 (7.17) | -0.8 (6.57)
  Change from Baseline to Month 6 (n=709,223) | -3.4 (7.64) | -0.6 (6.76)

10. Secondary Outcome: Physician-reported Clinical Global Impression of Improvement (CGI-I)
Description: The CGI-I is a rating scale allowing a physician-reported global evaluation of the subject's improvement over time. The Investigator assessed the subject's clinical change relative to the symptoms at baseline on the CGI-I, a seven-point scale, with rating as follows: 1=Very much improved, 2=Much improved, 3=Minimally improved, 4=No change, 5=Minimally worse, 6=Much worse, 7=Very much worse. The assessments were completed at Month 3 and Month 6. A lower score indicates improvement.
Time Frame: Month 3, Month 6
Population: This analysis was conducted using the Full Analysis Set. The Full Analysis Set comprised all randomized patients to whom study medication was assigned. Patients with month 3 and month 6 assessments were included in this analysis. Missing values were imputed using the Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatments (MS DMTs)
Number analyzed (Participants) | 789 | 263
units on a scale
  Month 3 (n=758,242) | 3.4 (1.02) | 3.9 (0.72)
  Month 6 (n=727,228) | 3.2 (1.11) | 3.9 (0.62)

ADVERSE EVENTS:
Description: In this analysis, patients with all (serious and non-serious) adverse events, serious adverse events and death were reported.
Groups:
- Standard MS DMT: Patients randomized in this arm received selected Standard MS DMT such as Interferon beta-1b or Interferon beta-1a or Glatiramer acetate for 6 months.
- Fingolimod Extension Phase: An open-label extension of up to 3 months of treatment with fingolimod was to be available for patients in the DMT arm who successfully completed all study visits.
Arm/Group | Fingolimod | Standard MS DMT | Fingolimod Extension Phase
Serious Adverse Events (participants affected / at risk) | 31/783 | 5/245 | 7/193
Other Adverse Events (participants affected / at risk) | 316/783 | 51/245 | 56/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=783) | Standard MS DMT (N=245) | Fingolimod Extension Phase (N=193)
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Basedow's disease (Endocrine disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Optic neuritis (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ileus (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Kidney infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 2 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 5 | 2 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=783) | Standard MS DMT (N=245) | Fingolimod Extension Phase (N=193)
Diarrhoea (Gastrointestinal disorders) | 41 | 4 | 3
Nausea (Gastrointestinal disorders) | 48 | 5 | 11
Fatigue (General disorders) | 90 | 14 | 10
Nasopharyngitis (Infections and infestations) | 43 | 13 | 7
Upper respiratory tract infection (Infections and infestations) | 51 | 8 | 9
Dizziness (Nervous system disorders) | 50 | 7 | 7
Headache (Nervous system disorders) | 97 | 8 | 19
Hypertension (Vascular disorders) | 43 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.